CLINICAL TRIAL: NCT00143741
Title: Use of Atorvastatin (Lipitor) to Decrease Panel Reactive Antibody Titers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atorvastatin 13815B
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: End-Stage Kidney Disease
Keywords: Kidney Disease, Lipitor, Atorvastatin, Allosensitization
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases | interventions — Atorvastatin

ARMS (1):
- Lipitor (Other)
  Interventions: Drug: Atorvastatin (Lipitor)

INTERVENTIONS:
Drug: Atorvastatin (Lipitor) — 20mg every day, taken by mouth. Dose could be increased up to 60mg every day during the course of the trial if tests indicate this is needed.

SUMMARY:
The purpose of this study is to identify subjects who are highly sensitized with antibodies. It is difficult for these patients to find suitable kidneys. We propose to treat such patients to decrease the antibodies in such a way, that it may become possible to safely transplant kidneys into them.

DETAILED DESCRIPTION:
Kidney transplantation is the desired treatment of choice in subjects with end-stage kidney disease (ESRD). The average waiting time for subjects to receive a "deceased donor" kidney transplant is 3-5 years. Currently, there are about 60,000 subjects on the national waiting list, and about 13,000-14,000 kidney transplants are performed each year. Approximately, 25% of subjects on the waiting list are "highly sensitized", meaning that they have natural proteins (antibodies) that aggressively protect their bodies from the invasion of foreign proteins. These individuals often have a difficult time accepting transplanted kidneys. The purpose of this study is to identify subjects who are highly sensitized with these antibodies, and treat them in such a way, that it may become possible to transplant kidneys into them. Drugs like atorvastatin (Lipitor) may decrease the levels of these anti-bodies and increase the possibility of these subjects to receive a kidney transplant. This research study is being done because currently, there are very limited and cumbersome treatment options to address this issue, subjects who are highly sensitized with antibodies, may unfortunately wait for a very long time or may never get transplanted.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years or older,
2. On the waiting list for a kidney transplant list
3. On hemodialysis or peritoneal dialysis

Exclusion Criteria:

1. Pregnant woman
2. Patients who need ongoing blood products
3. Patients with failed organs having active rejection
4. Other therapies to decrease PRA
5. Patients listed for multi-organ transplants (other than kidney-pancreas)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
This study is to identify subjects who are highly sensitized with these antibodies, and treat them in such a way, that it may become possible to transplant kidneys into them. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Kadambi, MD, Principal Investigator — The University of Chicago, 5841 South Maryland Ave., MC 5100 Chicago, IL 60637
Locations (1):
- The University of Chicago, Chicago, Illinois, United States